CLINICAL TRIAL: NCT04025931
Title: A Single-arm, Multi-center, Open, Phase II Study of Chidamide Combined With Toripalimab in Refractory and Advanced Soft-tissue Sarcoma
Brief Title: Chidamide Combined With Toripalimab in Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xing Zhang, Vice director of department of medical sarcoma and melanoma,Principal Investigator,Clinical Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SunYat-senU-chidamide
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chidamide combined with Toripalimab (Experimental): chidamide 30mg orally twice a week;
  240 mg of toripalimab (fixed dose) every three weeks.
  Repeat every three weeks. Patients with disease control (CR + PR + SD) and tolerable adverse reactions continued to take medication until the researchers concluded that patients were not suitable to continue medication or the efficacy evaluation was disease progression (PD). No other antineoplastic treatment can be given during the treatment.
  Interventions: Drug: chidamide and toripalimab

INTERVENTIONS:
Drug: chidamide and toripalimab — The eligible patients with advanced soft tissue sarcoma were treated with chidamide combined with toripalimb. Chidamide 30mg orally twice a week;
  Toripalimab 240 mg (fixed dose) every three weeks.
  Repeat every three weeks. Patients with disease control (CR + PR + SD) and tolerable adverse reactions continued to take medication until the researchers concluded that patients were not suitable to continue medication or the efficacy evaluation was disease progression (PD). No other antineoplastic treatment can be given during the treatment.

SUMMARY:
Soft tissue sarcoma is a relatively rare malignant tumor with an incidence of about 1-2/100,000. The best way to obtain evidence-based medical evidence is to participate in clinical trials with new drugs (especially targeted drugs and immunotherapy). Chidamide, an oral subtype-selective histone deacetylase inhibitor monotherapy was effective on the patients with hematological tumors by inhibiting HDAC activity and other ways, showing good anti-tumor activity. Histone deacetylase inhibitors (HDACi) may also reverse drug resistance or inefficiency of immunoassay inhibitors, and combination therapy has shown preliminary efficacy in a variety of tumors.Because of the poor prognosis of advanced soft tissue sarcoma, there is no standard second-line treatment. Therefore, we think it is necessary to explore the feasibility of combination of chidamide and Toripalimab monoclonal antibody in advanced, refractory and progressive soft tissue sarcoma after failure of standard treatment, and look forward to further improving the efficacy of soft tissue sarcoma.

DETAILED DESCRIPTION:
Histone deacetylase inhibitor (HDACI) can inhibit many kinds of hematological tumors by inhibiting HDAC activity and other ways, showing good anti-tumor activity. Chidamide is a new chemical structure benzamide HDAC inhibitor developed independently in China. It has the selectivity of HDAC subtypes and unique efficacy. In a phase II clinical study of Chidamide in the treatment of peripheral T-cell lymphoma in China in 2009, 79 patients with recurrent or refractory lymphoma had ORR of 27.9%. The 2016 edition of the Chinese Expert Consensus on Chidamide in the Treatment of PTCL discussed in detail the treatment of Chidamide alone or in combination with other drugs.

The representative drug of immunological checkpoint inhibitors is programmed death 1 (PD-1/PD-L1). PD-1/PD-L1 immunotherapy activates the body's own immune system to attack cancer cells by blocking the PD-1/PD-L1 pathway with drugs. Immunotherapy show its long-term control of cancer and its effectiveness in a variety of cancers.

In a multicenter phase II clinical trial, 80 patients with bone and soft tissue sarcoma were treated with single drug of PD-1 antibody Pembrolizumab. The results showed that all the patients with soft tissue sarcoma achieved therapeutic effect were undifferentiated pleomorphic sarcoma and liposarcoma. The overall objective remission rate was 18% (7/40), suggesting that Pembrolizumab alone does not fully activate suppressed T cells, and may need to be combined to improve the efficacy.

Recent studies have shown that combination of epigenetic regulators, such as histone deacetylase inhibitors (HDACi), can overcome some major drug resistance constraints and ensure patient safety. Pre-clinical data based on mouse models strongly support the feasibility and effectiveness of combination therapy. In vitro and in vivo studies, combined use of pan- or class I selective HDACi can benefit further. Chidamide is mainly targeted at subtypes 1, 2, 3 and 10 of HDAC class I and class II B. It has a regulatory effect on the abnormal epigenetic function of tumors. By inhibiting the related HDAC subtypes to increase the acetylation level of chromatin histone, chromatin remodeling is initiated, which changes the gene expression of multiple signal transduction pathways (i.e. epigenetic changes), thereby inhibiting the cell cycle of tumors, inducing apoptosis of tumors, and having overall regulatory activity on cellular immunity. Induction and enhancement of natural killer cells (NK) and antigen-specific cytotoxic T cells (CTL) mediated tumor killing. Chidamide can also enhance the mechanism of dendritic cells presenting and maturing tumor antigens, inhibiting regulatory T cells (Treg) and MDSC cells, and promote the anti-tumor immune function through regulating the micro-environment of tumor immunosuppression.

Because of the poor prognosis of advanced soft tissue sarcoma, there is no standard treatment for second-line treatment. Therefore, we think it is necessary to explore the feasibility of combination of chidamide and Toripalimab in advanced, refractory and progressive soft tissue sarcoma after failure of standard treatment, and look forward to further improving the efficacy of soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily participated in this study and signed the informed consent;
2. The pathology diagnosed with at least one measurable lesion according to RECIST 1.1 standard. The pathology includes synovial sarcoma, leiomyosarcoma, angiosarcoma, undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma, liposarcoma, fibrosarcoma, clear cell sarcoma, epithelioid sarcoma, malignant peripheral nerve sheath tumor, undifferentiated sarcoma, rhabdomyosarcoma, dermatofibrosareoma promberans, ewing's sarcoma /primary neural ectoderm tumors, desmoplastic small round cell tumor, inflammatory myofibroblastic sarcoma, malignant solitary fibroma. Except for chondrosarcoma, osteosarcoma, malignant mesothelioma, alveolar soft tissue sarcoma, gastrointestinal stromal tumor;
3. Advanced sarcoma patients with refractory or distant metastasis after failure of first-line standard therapy;
4. 14 ~ 70 years old; ECOG PS score: 0~1; Expected survival beyond 3 months;
5. Adequate organ and bone marrow function, no serious hematopoietic dysfunction or heart, lung, liver, kidney, thyroid dysfunction and immune deficiency (no blood transfusion, granulocyte colony stimulating factor or other medical support was received within 14 days before the use of the research drug):
6. Major organs functions should meet the following standards within 7 days before treatment:

   Blood routine examination standard (without blood transfusion within 14 days) :

   Hemoglobin (HB) ≥90g/L; The absolute value of neutrophils (ANC) ≥1.5×109/L; Platelet (PLT) ≥80 ×109/L.

   Biochemical examination shall meet the following standards:

   Total bilirubin (TBIL) ≤ 1.5 times ULN (Upper Limit Of Normal); alanine aminotransferase （ALT）and aspartate aminotransferase AST≤2.5 times ULN. If accompanied by liver metastasis, ALT and AST≤5 times ULN；Serum creatinine（Cr）≤1.5 times ULN or creatinine clearance rate (CCr)≥ 60ml/min； Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥ normal low limit (50%).
7. Thyrotropin (TSH) or free thyroxine (FT4) or free triiodothyronine (FT3) were all within the normal range (+10%).
8. Women of reproductive age should agree to use contraceptives (such as intrauterine devices, contraceptives or condoms) during and within 6 months after the study; Negative serum or urine pregnancy test within 7 days prior to study enrollment and must be non-lactating;
9. Men should agree to use contraceptives during and within 6 months after the study period.

Exclusion Criteria:

1. Patients who have previously used chidamide or other histone deacetylase inhibitors;
2. Previous treatment with immunological checkpoint inhibitors (PD-1, PD-L1, CTLA-4, etc.);
3. Other malignancies that have occurred or are present at the same time within 5 years, except for cured cancers including carcinoma in situ of the cervix, non-melanoma skin cancer and superficial bladder tumor [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor infiltrating basement membrane)];
4. Start the study of systemic anti-cancer therapy within 28 days before treatment, including chemotherapy, immunotherapy, biotherapy (cancer vaccine, cytokines, or growth factors that control cancer).
5. The patients received Chinese herbal medicine or Chinese patent medicine treatment within 7 days before the start of the study.
6. Systemic anti-tumor therapy, including cytotoxic therapy, signal transduction inhibitors, and immunotherapy (or mitomycin C administration within 6 weeks before the treatment with the experimental drug), is planned within 4 weeks before enrollment or during the medication period of this study. In the first 4 weeks of enrollment, the patients were treated with field expanding radiotherapy (ef-rt) or the limited field radiotherapy designed to evaluate tumor lesions in the first 2 weeks of enrollment.
7. Accompanied by pleural effusion or ascites, causing respiratory syndrome (CTCAE grade 2 dyspnea [grade 2 dyspnea refers to shortness of breath when there is a small amount of activity; it affects instrumental daily life activities]);
8. Unrelieved toxic reactions caused by any previous treatment higher than CTCAE (4.1) level 1 or above, excluding hair loss;
9. Patients with brain metastases with symptoms or with symptoms for less than 2 months;
10. Patients with any severe and/or uncontrolled disease, including:

1)Patients with unsatisfactory blood pressure control (systolic blood pressure 150 mmHg, diastolic blood pressure 100 mmHg); 2)Patients with grade I or above myocardial ischemia or myocardial infarction, arrhythmia (including QTC 480ms) and grade II congestive heart failure (NYHA classification); 3)Active or uncontrolled severe infection (CTCAE grade 2 infection); 4)Cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatment; 5) Renal failure requires hemodialysis or peritoneal dialysis; 6) Have a history of immunodeficiency, including HIV positive or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation; 7)Poor control of diabetes mellitus (FBG) > 10mmol/L); 8)Urine routine test indicated urine protein ++, and confirmed the 24-hour urine protein quantitative > 1.0g; 9)Patients with seizures requiring treatment;

11. Received major surgical treatment, open biopsy or obvious traumatic injury within 28 days before enrollment;

12. Patients with any signs of bleeding constitution or medical history, regardless of the severity; Patients with any bleeding or bleeding event CTCAE level 3 within 4 weeks before enrollment have unhealed wounds, ulcers or fractures;

13. Hyperactive/venous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attack), deep venous thrombosis and pulmonary embolism;

14. Patients with active ulcer, intestinal perforation and intestinal obstruction;

15. Have a history of mental drug abuse and cannot quit or have mental disorder;

16. Participated in clinical trials of other anti-tumor drugs within 28 days before enrollment;

17.According to the judgment of the researcher, there are those who seriously endanger the safety of patients or affect the patients' completion of the study.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-01-19 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Objective response rate is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.

SECONDARY OUTCOMES:
Progress free survival | until Progressive Disease(PD) or death(up to 24 months)
  Progress free survival defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Overall Survival | From randomization until death (up to 24 months)
  Overall survival is defined as the time until death due to any cause.
Disease Control Rate | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-Sen Univerisity, Guangzhou, Guangdong, China